CLINICAL TRIAL: NCT00662467
Title: Warfarin After Anterior ST-Elevation Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Dr. J-D Schwalm, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-281
Record Dates: First submitted 2008-04-08; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Hemorrhage; Thromboembolism; Clopidogrel; Aspirin; Warfarin
MeSH Terms: conditions — Myocardial Infarction; Hemorrhage; Thromboembolism | interventions — Aspirin; Clopidogrel; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): aspirin and clopidogrel
  Interventions: Drug: aspirin + clopidogrel
- 2 (Experimental): aspirin, clopidogrel, and warfarin
  Interventions: Drug: aspirin + clopidogrel + warfarin

INTERVENTIONS:
Drug: aspirin + clopidogrel — Dual therapy
  Arms: 1
Drug: aspirin + clopidogrel + warfarin — Triple therapy
  Arms: 2

SUMMARY:
Following severe heart attacks involving the front wall of the heart (anterior myocardial infarction), patients are at risk of developing blood clots in the main pumping chamber that can cause a stroke. In the past, studies have shown that a blood thinner (warfarin) can decrease the risk of stroke and clot formation if administered to patients after an anterior myocardial infarction.

However, in today's current practice, certain heart attack patients are commonly treated with two blood-thinning medications (aspirin and clopidogrel) to prevent recurrent heart attacks.

Thus, a clinical problem is created as physicians are not clear how to treat patients after an anterior myocardial infarction who are at risk of a clot but require aspirin and clopidogrel to keep their blood vessels open. Adding warfarin to the combination of aspirin and clopidogrel will possibly decrease the risk of stroke but increase the risk of bleeding. Currently, there is no good evidence to help guide physicians. As demonstrated by a survey done at the Hamilton Health Sciences, there is a fifty/fifty split between physicians who use dual (aspirin and clopidogrel) versus triple (aspirin, clopidogrel, and warfarin) therapy in the treatment of similar patients as described above.

The purpose of this study is to address the bleeding and stroke complications in patients after a severe anterior myocardial infarction. Half of the eligible patients will receive dual therapy and half will receive triple therapy. We will compare the incidence of stroke, blood clots, and bleeding complications between the two groups at 3 months.

DETAILED DESCRIPTION:
Rationale:

Left ventricular mural thrombus (LVT) remains a common complication after anterior ST-elevation myocardial infarction (STEMI) with a reported incidence ranging from 12- 17%. Previous studies from the pre-thrombolytic era have shown that warfarin therapy significantly reduces the incidence of LVT and embolic events in patients post anterior STEMI. However, the risk/benefit ratio of warfarin therapy in the setting of early revascularization and dual antiplatelet therapy with aspirin and clopidogrel remains unknown.

Purpose:

To compare the incidence of death, MI, stroke, embolic events, LVT, and bleeding complications at 3 months in patients with an anterior STEMI and ejection fraction less than 40% treated with ASA and clopidogrel alone versus those treated with aspirin, clopidogrel, and warfarin (triple therapy group).

Sample Size:

This is a pilot project to help establish the feasibility of conducting a full scale externally funded study. As such sample size calculations are not applicable. The primary aim of the study is to determine the safety and feasibility of conducting a large-scale trial, and this pilot project in not expected to reveal a statistically significant difference between the 2 groups.

Design/Methodology:

All patients will be randomized to either aspirin and clopidogrel alone or to triple therapy with aspirin, clopidogrel and warfarin. The randomization process will be centralized and computer generated. Patients with a clear indication for oral anticoagulation such as atrial fibrillation, LV thrombus, mechanical heart valve, or DVT/PE will not undergo randomization but will be followed as part of a registry of patients on triple therapy. All patients will remain on the allocated therapy for 3 months at which time outcomes will be determined.

Study interventions:

Patients will be treated with either ASA and clopidogrel alone (dual therapy) or with aspirin, clopidogrel and warfarin (triple therapy) in combination for 3 months. Patients in the triple therapy arm will be bridged with intravenous unfractionated heparin, low molecular weight heparin, or fondaparinux until their INR is therapeutic, and will be followed by the thrombosis service for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Anterior STEMI
* An ejection fraction less than 40% as per initial LV angiography or echocardiogram
* Randomization possible within hospital admission if anticoagulated with no interruption > 24 hours
* Patient able and willing to give informed consent to participate in this trial

Exclusion Criteria:

* history of intracranial hemorrhage
* history of GI bleed last 6 months
* hemoglobin < 90 g/L
* platelet count < 100 x 10exp9/L
* ischemic stroke last 30 days
* intracranial tumor or aneurysm
* significant pericardial effusion
* severe renal failure (creatinine > 250 mmol/L).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Combined death, MI, embolic event (TIA, stroke, non-cns emboli), Major Bleeding, and LVT (as determined by echocardiography) at 3 months | 3 months

SECONDARY OUTCOMES:
Individual endpoints of LVT at discharge and at 3 months (determined by echocardiography), death, MI, stroke, TIA, non-CNS emboli, and minor bleeding | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jon-David R Schwalm, MD, FRCPC, Principal Investigator — McMaster University; Mayraj Ahmad, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences-Hamilton General Hopsital, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Nihoyannopoulos P, Smith GC, Maseri A, Foale RA. The natural history of left ventricular thrombus in myocardial infarction: a rationale in support of masterly inactivity. J Am Coll Cardiol. 1989 Oct;14(4):903-11. doi: 10.1016/0735-1097(89)90463-4. PMID 2794276
- [Background] Asinger RW, Mikell FL, Elsperger J, Hodges M. Incidence of left-ventricular thrombosis after acute transmural myocardial infarction. Serial evaluation by two-dimensional echocardiography. N Engl J Med. 1981 Aug 6;305(6):297-302. doi: 10.1056/NEJM198108063050601. PMID 7242633
- [Background] Meltzer RS, Visser CA, Fuster V. Intracardiac thrombi and systemic embolization. Ann Intern Med. 1986 May;104(5):689-98. doi: 10.7326/0003-4819-104-5-689. PMID 3516044
- [Background] Kupper AJ, Verheugt FW, Peels CH, Galema TW, Roos JP. Left ventricular thrombus incidence and behavior studied by serial two-dimensional echocardiography in acute anterior myocardial infarction: left ventricular wall motion, systemic embolism and oral anticoagulation. J Am Coll Cardiol. 1989 Jun;13(7):1514-20. doi: 10.1016/0735-1097(89)90341-0. PMID 2723267
- [Background] Chiarella F, Santoro E, Domenicucci S, Maggioni A, Vecchio C. Predischarge two-dimensional echocardiographic evaluation of left ventricular thrombosis after acute myocardial infarction in the GISSI-3 study. Am J Cardiol. 1998 Apr 1;81(7):822-7. doi: 10.1016/s0002-9149(98)00003-4. PMID 9555769
- [Background] Nayak D, Aronow WS, Sukhija R, McClung JA, Monsen CE, Belkin RN. Comparison of frequency of left ventricular thrombi in patients with anterior wall versus non-anterior wall acute myocardial infarction treated with antithrombotic and antiplatelet therapy with or without coronary revascularization. Am J Cardiol. 2004 Jun 15;93(12):1529-30. doi: 10.1016/j.amjcard.2004.02.066. PMID 15194027
- [Background] Stratton JR, Lighty GW Jr, Pearlman AS, Ritchie JL. Detection of left ventricular thrombus by two-dimensional echocardiography: sensitivity, specificity, and causes of uncertainty. Circulation. 1982 Jul;66(1):156-66. doi: 10.1161/01.cir.66.1.156. PMID 7083502
- [Background] Vaitkus PT, Barnathan ES. Embolic potential, prevention and management of mural thrombus complicating anterior myocardial infarction: a meta-analysis. J Am Coll Cardiol. 1993 Oct;22(4):1004-9. doi: 10.1016/0735-1097(93)90409-t. PMID 8409034
- [Background] Weinreich DJ, Burke JF, Pauletto FJ. Left ventricular mural thrombi complicating acute myocardial infarction. Long-term follow-up with serial echocardiography. Ann Intern Med. 1984 Jun;100(6):789-94. doi: 10.7326/0003-4819-100-6-789. PMID 6721297
- [Background] Chen ZM, Jiang LX, Chen YP, Xie JX, Pan HC, Peto R, Collins R, Liu LS; COMMIT (ClOpidogrel and Metoprolol in Myocardial Infarction Trial) collaborative group. Addition of clopidogrel to aspirin in 45,852 patients with acute myocardial infarction: randomised placebo-controlled trial. Lancet. 2005 Nov 5;366(9497):1607-21. doi: 10.1016/S0140-6736(05)67660-X. PMID 16271642
- [Background] Sabatine MS, Blake GJ, Drazner MH, Morrow DA, Scirica BM, Murphy SA, McCabe CH, Weintraub WS, Gibson CM, Cannon CP. Influence of race on death and ischemic complications in patients with non-ST-elevation acute coronary syndromes despite modern, protocol-guided treatment. Circulation. 2005 Mar 15;111(10):1217-24. doi: 10.1161/01.CIR.0000157733.50479.B9. PMID 15769761
- [Background] Antman EM, Anbe DT, Armstrong PW, Bates ER, Green LA, Hand M, Hochman JS, Krumholz HM, Kushner FG, Lamas GA, Mullany CJ, Ornato JP, Pearle DL, Sloan MA, Smith SC Jr, Alpert JS, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Gregoratos G, Halperin JL, Hiratzka LF, Hunt SA, Jacobs AK; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; Canadian Cardiovascular Society. ACC/AHA guidelines for the management of patients with ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Revise the 1999 Guidelines for the Management of Patients with Acute Myocardial Infarction). Circulation. 2004 Aug 31;110(9):e82-292. No abstract available. PMID 15339869